CLINICAL TRIAL: NCT01716741
Title: Identification of Undiagnosed Gaucher Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Michael Murray, Clinical Chief, Division of Genetics, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P000469
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-08

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; lysosomal storage disorder; metabolic disease; medical records review
MeSH Terms: conditions — Gaucher Disease; Lysosomal Storage Diseases; Metabolic Diseases | interventions — Restriction Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzyme analysis (Other): Patients invited for evaluation will undergo glucocerebrosidase enzyme analysis
  Interventions: Other: Enzyme analysis

INTERVENTIONS:
Other: Enzyme analysis

SUMMARY:
Partners HealthCare maintains a Patient Data Registry (PDR) with information from all patient encounters at Partners HealthCare facilities. We intend to utilize the PDR to identify groups of patient who are of high clinical suspicion for undiagnosed Gaucher disease. A group of potential participants will be identified through the PDR. Detailed records will be requested to further narrow to ideal participants based upon previously existing diagnoses and symptoms. Participants will be invited to partake in the study via a letter from their Partners care provider with supporting study details. Study participants will be evaluated in a one-time visit. A complete family and medical history will be collected. A physical exam will be performed, and up to 20cc of blood will be drawn. All participants will be notified of their disease status via letter and phone call from the study staff. If the study participant is diagnosed with GD through this evaluation, proper follow-up recommendations and referrals will be provided. Our intent is to determine if existing patient data can successfully be utilized to aid in the identification of patients with rare genetic disease.

ELIGIBILITY:
Inclusion Criteria:

* Must have records available in the Partners HealthCare Patient Data Registry

Exclusion Criteria:

* Must not have a diagnosis of Gaucher disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
number of patients with previously undiagnosed GD identified | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Murray, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hosptial, Boston, Massachusetts, United States